CLINICAL TRIAL: NCT04534374
Title: Acute Multiple Joint, Structural Barbell Resistance Exercise Improves Information Processing Speed and Decreases Conflict-related Neural Activity in Older Adults: A Crossover, Sham Control, Randomized Control Trial With REP
Brief Title: Multiple Joint, Structural Barbell Resistance Exercise Improves Information Processing Speed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Ting-Yu Lin, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201807HM004
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Decline; Aging
Keywords: exercise; resistance training; kinesiology; cognition; ERP; neuroimage
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise (Experimental): The experimental intervention is a session of resistance exercise described in the intervention section.
  Interventions: Behavioral: Resistance exercise
- Stretching exercise (Active Comparator): The active control intervention is a session of stretching exercise described in the intervention section.
  Interventions: Behavioral: Stretching exercise (sham exercise)

INTERVENTIONS:
Behavioral: Resistance exercise — Barbell back squat, press, and deadlift for three sets of five repetitions with the weight closest to 75% of their estimated 1 repetition max. The participants were instructed to execute the movement with moderate speed (2s eccentric, 2s concentric, no pause in between). The rest period between sets and exercise movements was two to three minutes.
  Arms: Resistance exercise
Behavioral: Stretching exercise (sham exercise) — Participants completed a passive stretching exercise session for a similar duration of time as the resistance exercise (≈ 30 min) as sham intervention, which included 15-20 stretching movements twice, holding each for 30 seconds as recommended by ACSM.
  Arms: Stretching exercise

SUMMARY:
This study investigated the effect of acute multiple joint, structural barbell resistance exercise on information processing speed and conflict-related neural activity in older adults via a crossover, sham control, randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. male adults aged 50-65 years old
2. exercise ≥ 150 minutes/week
3. normal or corrected-to-normal vision
4. right-handed

Exclusion Criteria:

1. dementia (MMSE ≥ 24)
2. any medical condition listed on PARQ
3. depression (BDI-II score ≤ 13)
4. any diagnostic cardiovascular, neurological and other chronic diseases

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change of Information processing speed between resistance and stretching exercises | 5-30 minutes before and 10-35 minutes after each intervention.
  Choice reaction time of the Stroop test congruent condition. Unit: millisecond. Shorter reaction time means a better outcome.
Change of Inhibitory control between resistance and stretching exercises | 5-30 minutes before and 10-35 minutes after each intervention.
  Interference score of the Stroop test. Unit: millisecond. Smaller interference score means a better outcome.

SECONDARY OUTCOMES:
Change of Conflict-related neural activity between resistance and stretching exercises | 5-30 minutes before and 10-35 minutes after each intervention.
  N2b (event-related potential)
Change of Neural activity related to locus coeruleus phasic response between resistance and stretching exercises | 5-30 minutes before and 10-35 minutes after each intervention.
  P3 (event-related potential)

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Min Hung, Ph.D., Study Chair — Department of Physical Education, National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The participant-level data and statistical code are available on request and the data will be anonymized.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Three years within the publication.

REFERENCES:
- [Derived] Lin TY, Hsieh SS, Chueh TY, Huang CJ, Hung TM. The effects of barbell resistance exercise on information processing speed and conflict-related ERP in older adults: a crossover randomized controlled trial. Sci Rep. 2021 Apr 28;11(1):9137. doi: 10.1038/s41598-021-88634-5. PMID 33911153